CLINICAL TRIAL: NCT01685814
Title: Lenalidomide, Adriamycin, Dexamethasone (RAD) Versus Lenalidomide, Bortezomib, Dexamethasone (VRD) for Induction in Newly Diagnosed Multiple Myeloma Followed by Response-adapted Consolidation and Lenalidomide Maintenance - A Randomized Multicenter Phase III Trial by Deutsche Studiengruppe Multiples Myelom (DSMM XIV
Brief Title: Lenalidomide, Adriamycin, Dexamethasone (RAD) Versus Lenalidomide, Bortezomib, Dexamethasone (VRD) for Induction in Newly Diagnosed Multiple Myeloma Followed by Response-adapted Consolidation and Lenalidomide Maintenance
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Wuerzburg University Hospital (Other)
Collaborators: ClinAssess GmbH (Industry); Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DSMM XIV; 2009-016616-21 (EudraCT Number)
Record Dates: First submitted 2012-06-27; First posted 2012-09-14 (Estimated); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Previously Untreated Symptomatic Multiple Myeloma
Keywords: multiple myeloma; autologous stem cell transplant; allogeneic stem cell transplant; lenalidomide; bortezomib
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- single stem cell transplant, 3-year lenalidomide maintenance (Active Comparator): Arm A
  Interventions: Drug: Lenalidomide, Bortezomib; Biological: autologous stem cell transplant
- tandem autologous transplant, lenalidomide maintenance (Experimental): Arm B
  Interventions: Drug: Lenalidomide, Bortezomib; Biological: autologous stem cell transplant
- allogeneic stem cell transplant, lenalidomide maintenance (Active Comparator): Arm C
  Interventions: Drug: Lenalidomide, Bortezomib; Biological: autologous stem cell transplant; Biological: allogeneic stem cell transplant
- tandem autologous transplant (Experimental): Arm D
  Interventions: Drug: Lenalidomide, Bortezomib; Biological: autologous stem cell transplant

INTERVENTIONS:
Drug: Lenalidomide, Bortezomib — Induction: two versus one novel drug maintenance: lenalidomide as a maintenance therapy
Biological: autologous stem cell transplant
Biological: allogeneic stem cell transplant
  Arms: allogeneic stem cell transplant, lenalidomide maintenance

SUMMARY:
The investigators propose this study utilizing Lenalidomide, Adriamycin, Dexamethasone (RAD) as comparator arm for Lenalidomide, Bortezomib, Dexamethasone (VRD) with the latter being considered a novel "standard" as an induction protocol, since response in general occurs early after starting treatment we decided to choose three cycles of either induction regimen.

Together with the "novel compounds", tandem high-dose melphalan is still the standard of care; it seems desirable to re-address the question of the number of transplant (single vs. double high-dose melphalan) procedures required in the context of triplet-induction protocols utilizing at least one of the novel compounds.

Thus, the question to be asked in the current protocol is whether immediate lenalidomide maintenance (i.e. following one cycle of high-dose therapy) as an investigational agent will result in identical progression free survival (PFS) when compared to tandem high-dose melphalan with deferred maintenance therapy.

Despite induction with novel compounds, approximately 25 - 40% of patients will be in less than very good partial response. Very recently, achievement of less than VGPR was confirmed to negatively impact on both PFS as well as overall survival (OS). Therefore, allogeneic stem cell transplantation is considered the standard of care in patients with suboptimal response to a first autograft.

In the current protocol, the standard for favourable responders (tandem-autologous transplant) is combined with 3 years of lenalidomide maintenance. This approach will be investigated for patients with less than VGPR following a first autotransplant and compared to the current standard of intensification in poor responders (allogeneic transplantation).

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent form
* Patients willing and able to undergo autologous and allogeneic transplantation
* no previous systemic therapy for the treatment of multiple myeloma (dexamethasone at a cumulative dose of 320 mg; plasmapheresis/dialysis without concomitant chemotherapy, local irradiation of bone lesions; and surgical intervention is accepted as pretreatment)
* Newly diagnosed multiple myeloma according to common diagnostic criteria including presence of CRAB and measurable disease parameters
* Cardiac ejection fraction (LVEF) of at least 50%
* Corrected DLCO of at least 50% ; alternatively pO2 [art.] of at least 70mmHg
* Karnofsky performance status of greater or equal to 50%
* adequate bone marrow function
* adequate serum chemistry values
* Use of adequate contraception for female subjects with childbearing potential and male subjects
* Bone marrow sample available for analysis of molecular cytogenetics
* Able to administer low molecular-weight heparin as a prophylactic anticoagulation therapy for the first three months(applicable for subjects randomized to RAD) and able to administer ASS 100 mg/d (applicable for subjects randomized to VRD)

Exclusion Criteria:

* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form
* Pregnant or lactating females
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk
* History of myocardial infarction; NYHA Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias; concomitant pericarditis or peri-/myocarditis
* Use of any other experimental drug or therapy within 28 days of baseline
* Greater or equal to Grade 2 peripheral neuropathy on clinical examination within 14 days before enrollment
* Known intolerance of boron
* Hypersensitivity to acyclovir or similar anti-viral drug
* Prior malignancy except adequately treated basal cell or squamous cell skin cancer, in situ cervical, breast or prostate cancer
* HIV positive, active hepatitis B, C or D viral infection, known CMV reactivation/active infection, EBV reactivation/active infection or treponema pallidum infection
* Uncontrolled diabetes mellitus
* Non-secretory MM
* Clinically relevant active infection or serious co-morbid medical conditions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Estimated)
Dates: Start 2012-05; Primary Completion 2016-09 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy endpoint for the induction phase is the rate of patients with CR at first restaging | within 8 days after end of last induction cycle ((Day 92(RAD); Day 71(VRD))
In the consolidation phase the primary efficacy endpoint for comparison II (response <VGPR after first ASCT) is the PFS rate | 3 years after the first ASCT, calculated from day 1 of ASCT.

SECONDARY OUTCOMES:
ORR following 3 cycles of induction treatment (VRD vs RAD) | within 8 days after end of last induction cycle
CR and ORR at the end of the whole treatment programme | at the end of the whole treatment programme (approx. 8 years)
Overall survival (OS) | 8 years from study entry
Incidence, severity and relationship of SAEs | 30 days post last dosing of study drug
Numbers of hospital stays and hospitalization days | within two years from second restaging

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Knop, MD, Study Director — Wuerzburg University Hospital; Hermann Einsele, MD, Principal Investigator — Wuerzburg University Hospital
Locations (32):
- Germany (32):
  - Universitätsklinikum Aachen, Med. Klinik IV, Hämatologie u. Onkologie, Aachen
  - Schön Klinik Starnberger See, Hämatologie und Onkologie, Berg
  - Charité Campus Virchow-Klinikum, Hämatologie, Onkologie u. Tumorimmunologie, Berlin
  - Klinikum Bremen-Mitte gGmbH, Klinik für Innere Medizin I, Bremen
  - Universitätsklinikum Carl Gustav Carus an der TU Dresden, Medizinische Klinik und Poliklinik I, Dresden
  - Universitätsklinikum Erlangen, Medizinische Klinik 5, Erlangen
  - Malteser Krankenhaus St. Franziskus-Hospital, medizinische Klinik I, Flensburg
  - Klinikum Frankfurt (Oder) GmbH Medizinische Klinik I, Frankfurt (Oder)
  - Klinikum der Johann Woflgang Goethe Universität, Frankfurt am Mai, Frankfurt am Main
  - Universitätsklinikum Freiburg, Abteilung für Innere Medizin I, Freiburg im Breisgau
  - Universitätmedizin Greifswald, Klinik und Poliklinik für Innere Medizin C, Greifswald
  - St. Marien-Hospital gem. GmbHKna, Hamm
  - Universitätsklinikum des Saarlandes Innere Medizin I, Homburg/Saar
  - Klinikum der Friedrich-Schiller-Universität Jena, Klinikum für Innrere Medizin II, Jena
  - Städtisches Klinikum Karlsruhe Medizinische Klinik III, Abt. Hämatologie u. Onkologie, Karlsruhe
  - Universitätsklinikum Schleswig-Holstein Campus Kiel, II. Med. Poliklinik, Kiel
  - Universitätsklinikum Schleswig-Holstein, Medizinische Klinik und Poliklinik II im städtischen Krankenhaus Kiel, Kiel
  - Stiftungsklinikum Mittelrhein GmbH, Klinik für Innere Medizin, Koblenz
  - Universitätsklinikum Schleswig-Holstein, Campus Lübeck, Medizinische Klinik I, Lübeck
  - Universitätsmedizin Mannheim medizinische Klinik III, Mannheim
  - Klinikum Schwabing, München
  - Klinikum der Universität München-Großhadern, München
  - III. Med. Klinik und Poliklinik, Klinikum rechts der Isar der TU München, München
  - Universitätsklinikum Münster, Medizinische Klinik u. Poliklinik A, Münster
  - Klinikum Nürnberg Nord, 5. Medizinische LKinik, Onkologie/Hämatologie, Nuremberg
  - Klinikum Oldenburg GmbH, Klinik für Innere Medizin II, Oldenburg
  - Uniklinikum Regensburg, Abteilung für Hämatologie und internistische Onkologie, Regensburg
  - Robert-Bosch-Krankenhaus, Abt. Hämatologie, Onkologie u. Palliativmedizin, Stuttgart
  - Universitätsklinikum Ulm,Klinik für Innere Medizin III, Ulm
  - Schwarzwald-Baar Klinkum Villingen-Schwennigen GmbH, Villingen-Schwenningen
  - Dr. Horst Schmidt Kliniken, Klinik Innere Medizin III, Wiesbaden
  - Universitätsklinikum Wuerzburg, Medizinische Klinik II, Würzburg